CLINICAL TRIAL: NCT04276207
Title: Effects of LY900014 on Recovery From Hyperglycemia Compared to Humalog in Subjects With Type 1 Diabetes Mellitus (T1DM) on Continuous Subcutaneous Insulin Infusion
Brief Title: A Study of LY900014 Versus Insulin Lispro (Humalog) on High Blood Sugar in Participants With Type 1 Diabetes Who Use Insulin Pumps
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 17277; I8B-MC-ITST (Other: Eli Lilly and Company); 2019-003493-13 (EudraCT Number)
Record Dates: First submitted 2020-02-18; First posted 2020-02-19 (Actual); Results first posted 2021-08-25 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-07

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Lispro

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- 100 U/mL LY900014 (Experimental): 100 units per milliliter (U/mL) LY900014 administered by continuous subcutaneous insulin infusion (CSII) in one of two study periods.
  Interventions: Drug: LY900014
- 100 U/mL Insulin Lispro (Humalog) (Active Comparator): 100 U/mL Insulin Lispro (Humalog) administered by CSII in one of two study periods.
  Interventions: Drug: Insulin Lispro

INTERVENTIONS:
Drug: LY900014 — Administered by CSII
  Arms: 100 U/mL LY900014
Drug: Insulin Lispro — Administered by CSII
  Other Names: Humalog; LY275585
  Arms: 100 U/mL Insulin Lispro (Humalog)

SUMMARY:
The main purpose of this study is to compare LY900014 to insulin lispro (Humalog) in participants with type 1 diabetes who are using an insulin pump and have high blood sugar after eating. For each participant, the study will last about two to nine weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants with type 1 diabetes
* Body mass index (BMI) between 18.5 and 30.0 kilograms per square meter, inclusive
* Hemoglobin A1c (HbA1c) less than or equal to 8.5 percent (%)
* Using CSII and stable insulin regimen for at least 3 months prior to inclusion into the trial

Exclusion Criteria:

* Known or suspected hypersensitivity to investigational medical product(s) or related products
* Receipt of any medicinal product in clinical development within 30 days or at least 5 half-lives of the related substances and their metabolites (whichever is longer) before randomization in this trial
* Known slowing of gastric emptying and or gastrointestinal surgery that, in the opinion of the investigator, might change gastrointestinal motility and food absorption
* Proliferative retinopathy or maculopathy as judged by the Investigator based on a recent (less than 1.5 years) ophthalmologic examination
* Widespread subcutaneous lipodystrophy in the abdomen
* Current use of any glucose-lowering agents other than insulin within 3 months prior to screening
* Chronic or recent use of corticosteroids

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2020-02-25 (Actual); Primary Completion 2020-08-10 (Actual); Study Completion 2020-08-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Profil Mainz GmbH & Co. KG, Mainz, Rhineland-Palatinate, Germany

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Sequence AB (LY900014, Insulin Lispro (Humalog)): Period 1:
  Participants received 100 units per milliliter (U/mL) of LY900014 administered by continuous subcutaneous insulin infusion (CSII).
  Period 2:
  Participants received 100 U/mL of Insulin lispro Humalog) administered by CSII.
- Sequence BA (Insulin Lispro (Humalog), LY900014)): Period 1:
  Participants received 100 U/mL of Insulin lispro (Humalog) administered by CSII.
  Period 2:
  Participants received 100 U/mL of LY900014 administered by CSII.
Period: Period 1
Arm/Group | Sequence AB (LY900014, Insulin Lispro (Humalog)) | Sequence BA (Insulin Lispro (Humalog), LY900014))
Started | 15 | 17
Received at Least One Dose of Study Drug | 15 | 17
Completed | 15 | 16
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Washout (3- 14 Days)
Arm/Group | Sequence AB (LY900014, Insulin Lispro (Humalog)) | Sequence BA (Insulin Lispro (Humalog), LY900014))
Started | 15 | 16
Completed | 15 | 16
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Sequence AB (LY900014, Insulin Lispro (Humalog)) | Sequence BA (Insulin Lispro (Humalog), LY900014))
Started | 15 | 16
Completed | 15 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- 100 U/mL LY900014 and 100 U/mL Insulin Lispro (Humalog): Participants received 100 U/mL LY900014 administered by CSII in one of two study periods.
  Participants received 100 U/mL Insulin Lispro (Humalog) administered by CSII in one of two study periods.
Arm/Group | 100 U/mL LY900014 and 100 U/mL Insulin Lispro (Humalog)
Number analyzed (Participants) | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.8 (9.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 32
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Germany | 32

OUTCOME MEASURES:

1. Primary Outcome: Time to Recovery From Hyperglycemia Following Administration of LY900014 and Insulin Lispro (Humalog) After Missed Meal Bolus
Description: Time to Recovery from Hyperglycemia was defined as tPG140 = time to achieve glucose of 140 Milligrams per deciliter (mg/dL).
Time Frame: Day 1: Baseline up to 5 hours after missed meal bolus
Population: All participants who received both study treatments with the same insulin dose and achieved recovery from hyperglycemia on day 1
Measure: Median (Full Range); unit: Hours
Groups:
- 100 U/mL LY900014: Participants received 100 U/mL of LY900014 administered by CSII in one of the two study periods.
- 100 U/mL Insulin Lispro (Humalog): Participants received 100 U/mL of Insulin lispro (Humalog) administered by CSII in one of the two study periods.
Arm/Group | 100 U/mL LY900014 | 100 U/mL Insulin Lispro (Humalog)
Number analyzed (Participants) | 21 | 21
Hours | 1.79 [0.85 to 4.25] | 2.55 [0.92 to 4.68]
Statistical Analysis 1: Comparison: 100 U/mL LY900014 vs 100 U/mL Insulin Lispro (Humalog); Test type: Superiority; p = 0.1450, Mixed Models Analysis; Mean Difference (Final Values) = -0.377, 95% CI 2-sided [-0.896 to 0.142]

2. Primary Outcome: Time to Recovery From Hyperglycemia Following Administration of LY900014 and Insulin Lispro (Humalog) After Pump Suspension
Description: Time to Recovery from Hyperglycemia was defined as tPG140 = time to achieve glucose of 140 mg/dL.
Time Frame: Day 2: Baseline up to 5 hours after pump suspension
Population: All participants who received both study treatments with the same insulin dose and achieved recovery from hyperglycemia on day 2
Measure: Median (Full Range); unit: Hours
Arm/Group | 100 U/mL LY900014 | 100 U/mL Insulin Lispro (Humalog)
Number analyzed (Participants) | 28 | 28
Hours | 1.53 [0.97 to 2.24] | 1.78 [1.33 to 2.44]
Statistical Analysis 1: Comparison: 100 U/mL LY900014 vs 100 U/mL Insulin Lispro (Humalog); Test type: Superiority; p = 0.0010, Mixed Models Analysis; Mean Difference (Final Values) = -0.262, 95% CI 2-sided [-0.406 to -0.117]

3. Secondary Outcome: Pharmacodynamics (PD): Maximum Observed Plasma Glucose (PGmax) Following Administration of LY900014 and Insulin Lispro (Humalog)
Description: PD: PGmax following administration of LY900014 and insulin lispro (Humalog)
Time Frame: Day 1: Baseline up to 5 hours after missed meal bolus and Day 2: Baseline up to 5 hours after pump suspension
Population: All participants who received both study treatments with the same insulin dose and achieved recovery from hyperglycemia on days 1 and 2
Measure: Mean (Standard Deviation); unit: Milligrams per deciliter (mg/dL)
Arm/Group | 100 U/mL LY900014 | 100 U/mL Insulin Lispro (Humalog)
Number analyzed (Participants) | 28 | 28
Milligrams per deciliter (mg/dL)
  Day 1: number analyzed (Participants) | 21 | 21
  Day 1 | 297 (27.6) | 309 (24.9)
  Day 2 | 259 (11.1) | 265 (9.26)
Statistical Analysis 1: Comparison: 100 U/mL LY900014 vs 100 U/mL Insulin Lispro (Humalog); Day 1; Test type: Superiority; p = 0.0173, Mixed Models Analysis; Mean Difference (Final Values) = -12.61, 95% CI 2-sided [-22.73 to -2.49]
Statistical Analysis 2: Comparison: 100 U/mL LY900014 vs 100 U/mL Insulin Lispro (Humalog); Day 2; Test type: Superiority; p = 0.0243, Mixed Models Analysis; Mean Difference (Final Values) = -5.75, 95% CI 2-sided [-10.69 to 0.81]

4. Secondary Outcome: Pharmacokinetics (PK): Time to Maximum Observed Insulin Lispro Concentration (Tmax) Following Administration of LY900014 and Insulin Lispro (Humalog)
Description: PK: Tmax following administration of LY900014 and insulin lispro (Humalog)
Time Frame: Day 1: Baseline up to 5 hours after missed meal bolus and Day 2: Baseline up to 5 hours after pump suspension
Population: as for outcome 3
Measure: Median (Full Range); unit: Hours
Arm/Group | 100 U/mL LY900014 | 100 U/mL Insulin Lispro (Humalog)
Number analyzed (Participants) | 28 | 28
Hours
  Day 1: number analyzed (Participants) | 21 | 21
  Day 1 | 0.75 [0.33 to 1.75] | 0.83 [0.33 to 1.75]
  Day 2 | 0.92 [0.25 to 2.25] | 0.92 [0.50 to 2.50]
Statistical Analysis 1: Comparison: 100 U/mL LY900014 vs 100 U/mL Insulin Lispro (Humalog); Day 1; Test type: Superiority; p = 0.945, Mixed Models Analysis
Statistical Analysis 2: Comparison: 100 U/mL LY900014 vs 100 U/mL Insulin Lispro (Humalog); Day 2; Test type: Superiority; p = 0.888, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: Baseline Up To 42 Days
Description: All randomized participants who received at least one dose of study drug.
Arm/Group | 100 U/mL LY900014 | 100 U/mL Insulin Lispro (Humalog)
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/32
Other Adverse Events (participants affected / at risk) | 3/31 | 2/32
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 100 U/mL LY900014 (N=31) | 100 U/mL Insulin Lispro (Humalog) (N=32)
Hyperglycaemia (Endocrine disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-01-22): https://cdn.clinicaltrials.gov/large-docs/07/NCT04276207/Prot_000.pdf
  • Statistical Analysis Plan (2020-07-15): https://cdn.clinicaltrials.gov/large-docs/07/NCT04276207/SAP_001.pdf